CLINICAL TRIAL: NCT02860000
Title: Randomized Phase II Trial to Evaluate Alisertib Alone or Combined With Fulvestrant for Women With Advanced, Endocrine-Resistant Breast Cancer
Brief Title: Alisertib With or Without Fulvestrant in Treating Patients With Locally Advanced or Metastatic, Endocrine-Resistant Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MC1431; NCI-2016-01211 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1431 (Other: Mayo Clinic); R01CA214893 (NIH); 15-000340 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2016-08-04; First posted 2016-08-09 (Estimated); Results first posted 2024-10-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Estrogen Receptor Status; HER2/Neu Negative; Invasive Breast Carcinoma; Postmenopausal; Stage III Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — MLN 8237; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (alisertib) (Experimental): Patients receive alisertib PO BID on days 1-3, 8-10, and 15-17. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression, may cross-over to Arm II.
  Interventions: Drug: Alisertib; Other: Laboratory Biomarker Analysis
- Arm II (alisertib, fulvestrant) (Experimental): Patients receive fulvestrant IM over 1-2 minutes on days 1 and 15 of course 1 and on day 1 of all subsequent courses. Patients also receive alisertib PO BID on days 1-3, 8-10, and 15-17. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alisertib; Drug: Fulvestrant; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Alisertib — Given PO
  Other Names: Aurora A Kinase Inhibitor MLN8237; MLN-8237; MLN8237
Drug: Fulvestrant — Given IM
  Other Names: Faslodex; Faslodex(ICI 182,780); ICI 182,780; ICI 182780; ZD9238
  Arms: Arm II (alisertib, fulvestrant)
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well alisertib with or without fulvestrant works in treating patients with endocrine-resistant breast cancer that has spread to other places in the body. Alisertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Hormone therapy using fulvestrant may fight breast cancer by blocking the use of estrogen by the tumor cells or reducing the amount of estrogen made by the body. Giving alisertib with or without fulvestrant may be better in treating patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the impact on objective tumor response rate (using Response Evaluation Criteria in Solid Tumors [RECIST] criteria) with the addition of fulvestrant to alisertib in women with endocrine resistant, advanced estrogen receptor positive breast cancer.

SECONDARY OBJECTIVES:

I. To evaluate the safety profile of each treatment regimen. II. To assess the impact on median progression-free survival with the addition of fulvestrant to alisertib.

III. To obtain estimated tumor response rate and the median progression-free survival time during alisertib and fulvestrant treatment in the cohort of patients who progress during alisertib monotherapy, and crossover to receive the combination of alisertib and fulvestrant.

TERTIARY OBJECTIVES:

I. To assess the changes in aurora A kinase, SMAD5 and SOX2 expression and phosphorylation in tumor tissue after first cycle of assigned treatment.

II. To assess the changes in estrogen receptor (ER) expression and function in tumor tissue after the first cycle of assigned treatment.

III. To generate patient derived xenografts (PDX) from tumors collected at baseline and progression of disease (PD) in order to identify mechanisms associated with both de novo and acquired alisertib resistance.

IV. After the first cycle of treatment, to assess changes in aurora A kinase, phosphorylated (p)~SOX2 and ER expression on circulating tumor cells (CTCs), and to assess concordance between change in expression with tumor tissue and CTCs.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive alisertib orally (PO) twice daily (BID) on days 1-3, 8-10, and 15-17. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression, may cross-over to Arm II.

ARM II: Patients receive fulvestrant intramuscularly (IM) over 1-2 minutes on days 1 and 15 of course 1 and on day 1 of all subsequent courses. Patients also receive alisertib PO BID on days 1-3, 8-10, and 15-17. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION ELIGIBILITY
* Post-menopausal defined as

  * Age >= 60 and amenorrhea > 12 consecutive months, OR
  * Age < 60 and amenorrhea > 12 consecutive months without another cause and documented follicle stimulating hormone (FSH) level of > 35 mIU/mL, OR
  * Previous bilateral oophorectomy
* Histologic proof of metastatic or locally advanced, unresectable breast cancer
* History of ER positive (+) (>= 10% of cells positive on hematoxylin and eosin stain [H&E]), HER2 negative (-) breast cancer disease, either as a

  * History of primary, operable ER+/HER2- invasive breast cancer OR
  * History of de novo metastatic breast cancer that is ER+/HER2-

    * Note: HER2- (negative) disease defined as one of the following:

      * HER2 immunohistochemistry (IHC) expression of 0, 1+ and in-situ hybridization (ISH) non-amplified
      * HER2 IHC expression of 0, 1+ and ISH not done
      * HER2 IHC expression of 2+ and ISH non-amplified
      * IHC not done and ISH non-amplified
* Prior treatment

  * No more than two prior chemotherapy regimens in the metastatic setting
  * Prior treatment with fulvestrant in the metastatic setting is required, except for patients with a history of ER-negative metastatic breast cancer
  * Unlimited prior endocrine therapy regimens in the metastatic setting are allowed
  * No prior treatment with an aurora Kinase inhibitor (either an aurora A or pan-aurora kinase inhibitor)
* Disease that is measurable where:

  * A non-nodal lesion is considered measurable if its longest diameter can be accurately measured as >= 2.0 cm with chest x-ray, or as >= 1.0 cm with computed tomography (CT) scan, CT component of a positron emission tomography (PET)/CT, or magnetic resonance imaging (MRI)
  * A malignant lymph node is considered measurable if its short axis is >= 1.5 cm when assessed by CT scan (CT scan slice thickness recommended to be no greater than 5 mm); Note: tumor lesions in a previously irradiated area are not considered measurable disease; Note: disease that is measurable by physical examination only is not eligible
* No history of tumors involving spinal cord or heart
* History of brain metastases as per the following criteria:

  * Patients with a history of resected brain metastases are eligible only if they are asymptomatic and have stable MRI scans for 3 consecutive months, including < 28 days prior to pre-registration
  * Patients who receive stereotactic radiosurgery or whole brain radiation for brain metastases are eligible only if they are asymptomatic and have stable MRI scans for 3 consecutive months, including < 28 days prior to pre-registration
* Fully recovered from acute, reversible effects of prior therapy regardless of interval since last treatment;

  * EXCEPTION: neuropathies - if grade 2 neuropathies have been stable for at least 3 months since completion of prior treatment patient is eligible
* Eastern Cooperative Oncology Group (ECOG) performance status: 0, 1, 2
* Not receiving administration of proton pump inhibitor, H2 antagonist, or pancreatic enzymes
* Willing to limit daily alcohol intake to the following: one 12-oz glass of beer, one 6-oz glass of wine, or one 1.5-oz portion of 80-proof alcohol
* No uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Uncontrolled symptomatic cardiac arrhythmia
  * Uncontrolled hypertension (defined as blood pressure > 160/90)
* No history of uncontrolled sleep apnea syndrome and other conditions that could result in excessive daytime sleepiness, such as severe chronic obstructive pulmonary disease; requirement for supplemental oxygen
* No other active second malignancy other than non-melanoma skin cancers and in situ cervical cancers within 5 years of registration

  * NOTE: A second malignancy is not considered active if all treatment for that malignancy is completed and the patient has been disease-free for at least 5 years prior to registration
* Ability to provide written informed consent
* Willing to return to enrolling institution for follow-up during the active treatment; event monitoring following completion of therapy may occur outside the enrolling institution
* No history of myocardial infarction =< 6 months prior to pre-registration or New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* No prior allogeneic bone marrow or organ transplantation
* No known clinical finding or suspicion of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C
* No co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Able to swallow oral medication
* No known gastrointestinal (GI) disease or GI procedures that could interfere with the oral absorption or tolerance of alisertib; examples include, but are not limited to partial gastrectomy, history of small intestine surgery, and celiac disease
* No visceral crisis: Visceral crisis is not the mere presence of visceral metastases, but implies severe organ dysfunction as assessed by symptoms and signs, laboratory studies, and rapid progression of disease
* No requirement for constant administration of proton pump inhibitor, H2 antagonist, or pancreatic enzymes
* Willing to undergo a biopsy of a metastatic site of breast disease for central laboratory determination of ER and correlative research purposes
* REGISTRATION ELIGIBILITY CRITERIA
* =< 28 days post pre-registration
* Central ER determination on pre-registration biopsy completed
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 9.0 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Alanine transaminase (ALT) =< 3 x ULN (=< 5 x ULN for patients with liver involvement)
* Calculated creatinine clearance must be >= 45 ml/min using the Cockcroft-Gault formula
* Willing to provide blood and tissue for correlative research purposes

Exclusion Criteria:

* REGISTRATION EXCLUSION CRITERIA
* Any of the following therapies prior to registration:

  * Chemotherapy =< 21 days
  * Immunotherapy =< 21 days
  * Biologic therapy =< 21 days
  * Hormonal therapy =< 14 days
  * Monoclonal antibodies =< 14 days
  * Radiation therapy =< 14 days
* Administration of myeloid growth factors or platelet transfusion =< 14 days prior to registration
* Systemic infection requiring intravenous (IV) antibiotic therapy =< 14 days prior to registration
* Treatment with clinically significant enzyme inducers, such as the enzyme-inducing antiepileptic drugs phenytoin, carbamazepine or phenobarbital, or rifampin, rifabutin, rifapentine or St. John's wort =< 14 days prior to registration
* Receipt of corticosteroids =< 7 days prior to registration, unless patient has been taking a continuous dose of no more than 15 mg/day of prednisone for at least 30 days prior to registration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tufia C. Haddad, M.D., Principal Investigator — Mayo Clinic
Locations (8):
- United States (8):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee

REFERENCES:
- [Derived] Haddad TC, Suman VJ, D'Assoro AB, Carter JM, Giridhar KV, McMenomy BP, Santo K, Mayer EL, Karuturi MS, Morikawa A, Marcom PK, Isaacs CJ, Oh SY, Clark AS, Mayer IA, Keyomarsi K, Hobday TJ, Peethambaram PP, O'Sullivan CC, Leon-Ferre RA, Liu MC, Ingle JN, Goetz MP. Evaluation of Alisertib Alone or Combined With Fulvestrant in Patients With Endocrine-Resistant Advanced Breast Cancer: The Phase 2 TBCRC041 Randomized Clinical Trial. JAMA Oncol. 2023 Jun 1;9(6):815-824. doi: 10.1001/jamaoncol.2022.7949. PMID 36892847
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Alisertib): Patients receive alisertib PO BID on days 1-3, 8-10, and 15-17. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression, may cross-over to Arm II.
  >
  > Alisertib: Given PO
  >
  > Laboratory Biomarker Analysis: Correlative studies
- Arm II (Alisertib, Fulvestrant): Patients receive fulvestrant IM over 1-2 minutes on days 1 and 15 of course 1 and on day 1 of all subsequent courses. Patients also receive alisertib PO BID on days 1-3, 8-10, and 15-17. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  >
  > Alisertib: Given PO
  >
  > Fulvestrant: Given IM
  >
  > Laboratory Biomarker Analysis: Correlative studies
Period: Initial Treatment
Arm/Group | Arm I (Alisertib) | Arm II (Alisertib, Fulvestrant)
Started | 47 | 49
Completed | 46 | 45
Not Completed | 1 | 4
Period: Optional Cross-over
Arm/Group | Arm I (Alisertib) | Arm II (Alisertib, Fulvestrant)
Started | 17 | 0
Completed | 17 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I (Alisertib): Patients receive alisertib PO BID on days 1-3, 8-10, and 15-17. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with disease progression, may cross-over to Arm II.> > Alisertib: Given PO>
  > Laboratory Biomarker Analysis: Correlative studies
- Arm II (Alisertib, Fulvestrant): Patients receive fulvestrant IM over 1-2 minutes on days 1 and 15 of course 1 and on day 1 of all subsequent courses. Patients also receive alisertib PO BID on days 1-3, 8-10, and 15-17. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.>
  > Alisertib: Given PO>
  > Fulvestrant: Given IM>
  > Laboratory Biomarker Analysis: Correlative studies
- Total: Total of all reporting groups
Arm/Group | Arm I (Alisertib) | Arm II (Alisertib, Fulvestrant) | Total
Number analyzed (Participants) | 46 | 45 | 91
Age, Customized [Count of Participants; unit: Participants]
  <40 (Years) | 3 | 4 | 7
  40-59 (Years) | 14 | 20 | 34
  60-74 (Years) | 25 | 19 | 44
  75+ (Years) | 4 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 45 | 91
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 45 | 41 | 86
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 41 | 39 | 80
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
BMI Group [Count of Participants; unit: Participants]
  Underweight | 0 | 1 | 1
  Normal | 14 | 21 | 35
  Overweight | 13 | 15 | 28
  Obese | 19 | 8 | 27
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG = 0: Fully active, able to carry on all pre-disease performance without restriction. > ECOG = 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work. > ECOG = 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours. > ECOG = 0 is better. ECOG = 2 is worse.
  Participants
    0 | 30 | 27 | 57
    1 | 16 | 18 | 34
Prior Taxane Based Therapy [Count of Participants; unit: Participants]
  No | 22 | 21 | 43
  Yes | 24 | 24 | 48
Prior Anthracycline Based Therapy [Count of Participants; unit: Participants]
  No | 29 | 23 | 52
  Yes | 17 | 22 | 39
Prior Capecitabine Regimen [Count of Participants; unit: Participants]
  No | 42 | 42 | 84
  Yes | 4 | 3 | 7
Prior Chemotherapy [Count of Participants; unit: Participants]
  No | 39 | 41 | 80
  Yes | 7 | 4 | 11
Prior Systemic Chemotherapy [Count of Participants; unit: Participants]
  No | 24 | 14 | 38
  Yes | 22 | 31 | 53
Prior Anastrozole Endocrine Therapy [Count of Participants; unit: Participants]
  No | 30 | 31 | 61
  Yes | 16 | 14 | 30
Prior Tamoxifen Treatment [Count of Participants; unit: Participants]
  No | 31 | 23 | 54
  Yes | 15 | 22 | 37
Prior Fulvestrant Treatment [Count of Participants; unit: Participants]
  No | 40 | 43 | 83
  Yes | 6 | 2 | 8
Prior Endocrine Therapy [Count of Participants; unit: Participants]
  No | 19 | 10 | 29
  Yes | 27 | 35 | 62
Prior Exemestane Therapy [Count of Participants; unit: Participants]
  No | 30 | 19 | 49
  Yes | 16 | 26 | 42
Prior Fulvestrant Therapy [Count of Participants; unit: Participants]
  No | 1 | 9 | 10
  Yes | 45 | 45 | 90
Prior Biologic Therapy [Count of Participants; unit: Participants]
  No | 27 | 27 | 54
  Yes | 19 | 18 | 37
Prior Everolimus Therapy [Count of Participants; unit: Participants]
  No | 29 | 19 | 48
  Yes | 17 | 26 | 43
Clinical Resistance to Endocrine Therapy [Count of Participants; unit: Participants] — Primary endocrine resistance- recurrence within the first 2 years of adjuvant endocrine therapy, or progression within the first 6 months of initiating first-line endocrine therapy for MBC Secondary endocrine resistance- recurrence during years 2-5 of adjuvant endocrine therapy (or within 12 months of completing adjuvant endocrine therapy) or progression occurring 6 or more months after initiating endocrine therapy for MBC.
  Participants
    Primary endocrine resistance | 11 | 8 | 19
    Secondary endocrine resistance | 35 | 37 | 72
ER findings from registration biopsy [Count of Participants; unit: Participants] — Immunofluorescent staining for selected markers (e.g., cytokeratins, EpCAM, DAPI, CD45, HER2, ER, Aurora A kinase, p-SMAD5, and p-SOX2) is used for the efficient positive and negative identification of CTCs via automated scanning digital microscopy and image analysis.
  Participants
    ER positive (>= 10% staining) | 40 | 39 | 79
    ER weakly positive (1 to 9.9% staining) or ER negative (0% staining) | 6 | 6 | 12
ER status [Count of Participants; unit: Participants] — Immunofluorescent staining for selected markers (e.g., cytokeratins, EpCAM, DAPI, CD45, HER2, ER, Aurora A kinase, p-SMAD5, and p-SOX2) is used for the efficient positive and negative identification of CTCs via automated scanning digital microscopy and image analysis.
  ER positive (≥ 10% staining) ER weakly positive (1 to 9.9% staining) or ER negative (0% staining)
  Participants
    Negative | 5 | 1 | 6
    Positive | 41 | 44 | 85
Bone Metastatic Disease [Count of Participants; unit: Participants]
  Yes | 40 | 39 | 79
  No | 6 | 6 | 12
Liver Metastatic Disease [Count of Participants; unit: Participants]
  Yes | 32 | 35 | 67
  No | 14 | 10 | 24
Nodal Metastatic Disease [Count of Participants; unit: Participants]
  Yes | 25 | 22 | 47
  No | 21 | 23 | 44

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate Defined as 100% Times the Number of Patients Who Meet the Criteria for Complete Response (CR) or Partial Response (PR) Using RECIST Criteria Version 1.1
Description: For arm I, tumor response rate is defined as 100% times the number of patients who meet the criteria for CR or PR on 2 consecutive evaluations approximately 8 weeks apart during treatment with alisertib monotherapy divided by the number of patients who started alisertib monotherapy. For arm II, tumor response rate is defined as 100% times the number of patients who meet the criteria for CR or PR on 2 consecutive evaluations approximately 8 weeks apart during treatment with combination of alisertib and fulvestrant divided by the number of patients who started treatment with the combination of a
Time Frame: Up to 4.5 years
Measure: Median (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm I (Alisertib) | Arm II (Alisertib, Fulvestrant)
Number analyzed (Participants) | 46 | 45
Percentage of Participants | 19.6 [10.6 to 31.7] | 29.9 [19.9 to 32.3]

2. Secondary Outcome: Biomarkers and ER Alpha Expression Assessed Using Tumor Tissue
Description: Spearman rank correlation coefficient will be used to examine the association between ER alpha expression and the biomarkers: CD44, CD24, total and phosphorylated expression of AURKA, SMAD5, and SOX2. A two sample test of the difference in proportions will be used to examine whether weak or no phosphorylated expression of AURKA, SMAD5, and SOX2 after one cycle of alisertib is associated with clinical benefit (CR + PR + stable disease on treatment for at least 6 months).
Time Frame: Up to 4 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Change in Blood Biomarker Levels
Description: Percent change in CTC expression of aurora A kinase, ER, and phospho- SOX2 expression from pre-treatment levels will be determined for each patient. Bland-Altman plots and weighted kappa statistics will be used to examine the concordance between the percent change in aurora A kinase, ER, and phospho-SOX2 expression from pre-treatment levels in CTC and in tumor tissue.
Time Frame: Baseline to 28 days
Reporting Status: Not Posted

4. Secondary Outcome: Change in Tumor Biomarker Levels
Description: Spearman rank correlation coefficient will be used to examine the association of maximum percentage of tumor shrinkage during treatment with the percent change after 1 cycle of treatment in aurora A Kinase (AAK) expressing cells, as well as percent changes after 1 cycle of treatment in tissue ER alpha, SMAD5, SOX2 expression and phosphorylation.
Time Frame: Baseline to 28 days
Reporting Status: Not Posted

5. Secondary Outcome: Clinical Benefit Rate (CBR) During Initial Treatment Defined as Percentage of Patients Who Completed 6 Courses of Treatment Without Documentation of Disease Progression
Description: For initial treatment in each arm, the CBR at 24 weeks will be defined as the proportion of patients who completed 6 cycles of treatment without documentation of disease progression. A 90% confidence interval for the CBR will be constructed using the Duffy-Santner approach to take into account the sequential nature of the study design.
Time Frame: At 24 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Alisertib) | Arm II (Alisertib, Fulvestrant)
Number analyzed (Participants) | 46 | 45
percentage of participants | 41.3 [29.0 to 54.5] | 28.9 [18.0 to 42.0]

6. Secondary Outcome: Duration of Response Defined as Time From Randomization to Disease Progression Among Those Patients Whose Disease Meets the RECIST Criteria for CR or PR on 2 Consecutive Evaluations Approximately 8 Weeks Apart During Initial Treatment
Description: Will be estimated using the Kaplan-Meier method.
Time Frame: Up to about 5 years
Measure: Median (Full Range); unit: days
Arm/Group | Arm I (Alisertib) | Arm II (Alisertib, Fulvestrant)
Number analyzed (Participants) | 46 | 45
days | 465 [113 to 1031] | 259.5 [53 to 1863]

7. Secondary Outcome: Incidence of Adverse Events Graded by Common Terminology Criteria-Criteria for Adverse Events (CTCAE) Version 4.0
Description: The CTCAE version 4.0 will be used to grade and assign attribution to each adverse event reported during initial treatment and crossover treatment separately.
Time Frame: Up to 30 days after last administration of study drug
Reporting Status: Not Posted

8. Secondary Outcome: Overall Survival
Description: Will be estimated using the Kaplan-Meier method.
Time Frame: Up to 5 years
Reporting Status: Not Posted

9. Secondary Outcome: Progression-free Survival
Description: Will be estimated using the Kaplan-Meier method.
Time Frame: Time from randomization to the first of these disease events: local/regional or distant breast recurrence, DCIS or invasive breast disease in contralateral breast, non-breast second primary, or death due to any cause, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Alisertib) | Arm II (Alisertib, Fulvestrant)
Number analyzed (Participants) | 46 | 45
months | 5.6 [3.9 to 10.0] | 5.4 [3.0 to 7.8]

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Arm I (Alisertib) | Arm II (Alisertib, Fulvestrant)
All-Cause Mortality (participants affected / at risk) | 2/46 | 1/48
Serious Adverse Events (participants affected / at risk) | 12/46 | 12/48
Other Adverse Events (participants affected / at risk) | 45/46 | 47/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Alisertib) (N=46) | Arm II (Alisertib, Fulvestrant) (N=48)
Anemia (Blood and lymphatic system disorders) | 4 (5) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 1 (2) | 0 (0)
Mitral valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (2) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Investigations - Other, specify (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (7) | 4 (4)
Platelet count decreased (Investigations) | 2 (2) | 2 (2)
White blood cell decreased (Investigations) | 1 (1) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (3)
Edema cerebral (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (2) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Alisertib) (N=46) | Arm II (Alisertib, Fulvestrant) (N=48)
Anemia (Blood and lymphatic system disorders) | 34 (310) | 30 (192)
Mitral valve disease (Cardiac disorders) | 1 (3) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (4) | 0 (0)
Blurred vision (Eye disorders) | 2 (6) | 0 (0)
Dry eye (Eye disorders) | 1 (2) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 2 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 23 (184) | 19 (119)
Dysphagia (Gastrointestinal disorders) | 1 (4) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (10) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (6) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (3) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 19 (59) | 15 (34)
Nausea (Gastrointestinal disorders) | 17 (80) | 22 (95)
Vomiting (Gastrointestinal disorders) | 6 (18) | 15 (46)
Edema face (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 1 (2)
Fatigue (General disorders) | 41 (365) | 40 (236)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 2 (2) | 5 (8)
Pain (General disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 1 (2) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (2)
Upper respiratory infection (Infections and infestations) | 2 (2) | 2 (3)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1) | 4 (10)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 6 (6)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (2) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (14) | 0 (0)
Investigations - Other, specify (Investigations) | 1 (11) | 0 (0)
Lymphocyte count decreased (Investigations) | 7 (80) | 13 (110)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 30 (169) | 29 (117)
Platelet count decreased (Investigations) | 15 (93) | 15 (140)
Weight loss (Investigations) | 0 (0) | 2 (7)
White blood cell decreased (Investigations) | 28 (189) | 29 (178)
Anorexia (Metabolism and nutrition disorders) | 19 (100) | 19 (46)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (8) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Hypersomnia (Nervous system disorders) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (3) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 2 (5) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (3)
Anxiety (Psychiatric disorders) | 1 (2) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 1 (3)
Depression (Psychiatric disorders) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (4) | 2 (5)
Acute kidney injury (Renal and urinary disorders) | 7 (59) | 1 (5)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (40) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (8) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 20 (244) | 21 (128)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (5) | 0 (0)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (4) | 2 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (20) | 6 (10)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (2)
Social circumstances - Other, specify (Social circumstances) | 1 (1) | 0 (0)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (18) | 4 (12)
Lymphedema (Vascular disorders) | 0 (0) | 2 (3)
Thromboembolic event (Vascular disorders) | 1 (40) | 3 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT02860000/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/00/NCT02860000/ICF_001.pdf